CLINICAL TRIAL: NCT03017222
Title: Therapeutic Efficacy of Ramosetron for Treatment of Established PONV After Laparoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4-2015-0435
Record Dates: First submitted 2017-01-01; First posted 2017-01-11 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2017-01

CONDITIONS: Abdominal Mass
MeSH Terms: interventions — Ondansetron; ramosetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ondansetron group (Active Comparator)
  Interventions: Drug: Ondansetron
- Ramosetron group (Experimental)
  Interventions: Drug: Ramosetron

INTERVENTIONS:
Drug: Ondansetron — Ondansetron also has been reported as effective prophylactic and therapeutic 5-HT3 receptor antagonist for the treatment of PONV. Ramosetron has been shown to have a very strong effect for preventing PONV in previous meta-analyses, but in recent report, its clinical significance may be questioned to request for additional study.
  Arms: Ondansetron group
Drug: Ramosetron — Ramosetron is a newly developed selective 5-HT3 (5 hydroxytryptamine 3) receptor antagonist with longer duration of action up to 48hours and higher receptor affinity, than its previously developed congeners, including ondansetron.
  Arms: Ramosetron group

SUMMARY:
Patients who had at least two risk factors of PONV (Postoperative nausea and vomiting) and underwent laparoscopic surgeries under general anesthesia were assessed for eligibility. Patients who developed PONV within the first 2 hours after anesthesia received intravenously, in a randomized double-blind manner, ondansetron 4 mg or ramosetron 0.3 mg. Patients were then observed for 24 hours after drug administration. The incidence of nausea and vomiting, severity of nausea, requirements for rescue antiemetic and adverse effects at 0-2 and 2-24 hours after drug administration were evaluated. The primary endpoint was the rate of patients exhibiting complete response, defined as no emesis and no further rescue antiemetic medication for 24 hours after drug administration.

ELIGIBILITY:
Inclusion Criteria:

* age 19-65 years
* patients undergoing elective laparoscopic surgery under inhalational anesthesia
* duration of surgery between 30 min to 4 h
* ASA (American Society of Anesthesiologists) physical status I or II, and patients who had at least two of these risk factors
* female gender, history of motion sickness (MS) or PONV, nonsmoking, and the use of postoperative opioids.

Exclusion Criteria:

* patients with history of being allergic to 5-HT3 receptor antagonist
* patients with history of anticancer chemotherapy
* chronic opioids use, alcohol abuse, or drug abuse
* patients who took antiemetic medication within 24 h before surgery, steroids within 24 h before surgery or 24 h after surgery
* presence of renal (serum Cr > 1.6 mg/dl)
* hepatic(liver enzymes more than 2 times normal value) insufficiency
* patients converted to open laparotomy
* patient who are pregnant or breast-feeding
* patient with borderline QTc(corrected QT interval) prolongation (> 430 ms for male, >450 ms for female)
* patient not able to understand the scoring of pain or express the degree of PONV.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-09-07; Primary Completion 2016-04-02 (Actual); Study Completion 2016-04-02 (Actual)

PRIMARY OUTCOMES:
ratio of complete response | 24 hours after administration of study drug
  complete response is defined as no retching or vomiting and no secondary rescue antiemetic administration

SECONDARY OUTCOMES:
incidence of nausea and vomiting | 24 hours after administration of study drug